CLINICAL TRIAL: NCT07229404
Title: A Combined Single- and Multiple-dose, Open-label, Randomized, 6 x 3 Crossover Study to Investigate the Relative Bioavailability, Safety and Tolerability of Elinzanetant (BAY 3427080) in Healthy Female Participants
Brief Title: A Study to Investigate Relative Bioavailability, Safety and Tolerability of Single- and Multiple-doses of Elinzanetant in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22790
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Vasomotor Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Treatments are administered in sequence of A-B-C
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 2 (Experimental): Treatments are administered in sequence of A-C-B
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 3 (Experimental): Treatments are administered in sequence of C-A-B
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 4 (Experimental): Treatments are administered in sequence of C-B-A
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 5 (Experimental): Treatments are administered in sequence of B-C-A
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 6 (Experimental): Treatments are administered in sequence of B-A-C
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — Elinzanetant (BAY 3427080), dosage 1
Drug: Treatment B — Elinzanetant (BAY 3427080), dosage 2
Drug: Treatment C — Elinzanetant (BAY 3427080), dosage 3

SUMMARY:
The aim of this study is to examine the relative bioavailability of elinzanetant when administered in new oral formulations (treatment B and C) after both single and multiple oral doses, compared to its administration in soft gel capsule form (treatment A).

Study details include:

An ambulatory screening visit within 4 weeks prior to first treatment. Participants will be admitted to the ward on Day -1 of each period. On Day 1, either treatment B or treatment C will be administered fasted in the evening, followed by blood sampling for a 24-hour pharmacokinetic (PK) profile.

On Day 2, the multiple dosing starts 3 hours after a standardized dinner in the evening.

After the last dosing on Day 7, a complete PK profile for 24 hours will be collected.

If there are no medical objections, participants will be discharged from the study ward on Day 9 in the morning for a washout-out period of at least 10 days (240 hours after last dosing, after period 1 and 2) or, in period 3, after the follow-up examination.

The total duration of the study will be approximately 10 to 12 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria

* Female participant between 18 to 65 years of age (inclusive), at the time of signing the informed consent form (ICF).
* Participant is overtly healthy as determined by the investigator (including assessment of medical history, physical examination, blood pressure (BP), pulse rate, 12-lead electrocardiogram (ECG), body temperature, and clinical laboratory).
* Body weight of at least 50 kg and body mass index (BMI) above or equal to 18.0 and below or equal to 32.0 kg/m² at screening.
* Signed informed consent as described in Section 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

* Diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study intervention(s) will not be normal.
* Known or suspected allergy or hypersensitivity to any study intervention (active substances or excipients of the preparations) to be used in the study - including e.g. non-investigational medicinal products, challenge agents, or rescue medication.
* Febrile illness within 2 weeks before the start of the first study intervention.
* History of clinically relevant seizures.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), Bilirubin, or gamma-glutamyl transferase (GGT) > 1.2 x upper limit of normal (ULN).
* Previous (within 30 days before first administration of study intervention) or concomitant participation in another clinical study with study intervention(s).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
AUC(0-24)md after multiple oral dosing 3 h after light dinner in the evening (treatments A, B, C) | From Day 0 to Day 8
Cmax,md and Cmin,,md after multiple oral dosing 3 h after light dinner in the evening (treatments A, B, C) | From Day 0 to Day 8

SECONDARY OUTCOMES:
AUC(0-24) after single dose in the evening under fasted condition (treatments A, B, C). | From Day 0 to Day 8
Cmax after single dose in the evening under fasted condition (treatments A, B, C). | From Day 0 to Day 8
Number and severity of treatment-emergent adverse events (TEAEs) after first study intervention until follow up | From first dosing up to Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.